CLINICAL TRIAL: NCT04338360
Title: Expanded Access to Convalescent Plasma for the Treatment of Patients With COVID-19
Status: Approved for marketing | Type: Expanded Access
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Joyner, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 20-003312
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: COVID-19 convalescent plasma — COVID-19 convalescent plasma

SUMMARY:
This expanded access program will provide access to investigational convalescent plasma for patients in acute care facilities infected with SARS-CoV-2 who have severe or life-threatening COVID-19, or who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening disease.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* Laboratory confirmed diagnosis of infection with SARS-CoV-2
* Admitted to an acute care facility for the treatment of COVID-19 complications
* Severe or life threatening COVID-19, or judged by the treating provider to be at high risk of progression to severe or life-threatening disease
* Informed consent provided by the patient or healthcare proxy

Severe COVID-19 is defined by one or more of the following:

* dyspnea
* respiratory frequency ≥ 30/min
* blood oxygen saturation ≤ 93%
* partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
* lung infiltrates > 50% within 24 to 48 hours

Life-threatening COVID-19 is defined as one or more of the following:

* respiratory failure
* septic shock
* multiple organ dysfunction or failure

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joyner, MD, Principal Investigator — Mayo Clinic
Locations (12):
- United States (12):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System in Austin, Austin, Minnesota
  - Mayo Clinic Health System in Cannon Falls, Cannon Falls, Minnesota
  - Mayo Clinic Health System in Lake City, Lake City, Minnesota
  - Mayo Clinic Health System in Mankato, Mankato, Minnesota
  - Mayo Clinic Health System in Owatonna, Owatonna, Minnesota
  - Mayo Clinic Health System in Red Wing, Red Wing, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- [Derived] Bruno KA, Wright RS, Culberson J, Wieczorek MA, Hodge DO, Johnson PW, Jimenez YA, Whelan ER, Malavet JM, Larson KF, Senefeld JW, Wiggins CC, Klassen SA, Ricci J, Sher T, Carter RE, Joyner MJ, Fairweather D, Jaffe AS. Cardiac troponin T elevation predicts mortality in hospitalized COVID-19 patients. Am Heart J Plus. 2025 Dec 2;61:100690. doi: 10.1016/j.ahjo.2025.100690. eCollection 2026 Jan. PMID 41446701
- [Derived] Bruno KA, Wright RS, Culberson J, Wieczorek MA, Hodge DO, Johnson PW, Jimenez YA, Whelan ER, Malavet JM, Larson KF, Senefeld JW, Wiggins CC, Klassen SA, Ricci J, Sher T, Carter RE, Joyner MJ, Fairweather D, Jaffe AS. Cardiac Troponin T Elevation Predicts Mortality in Hospitalized COVID-19 Patients. medRxiv [Preprint]. 2025 Jul 5:2025.07.03.25330855. doi: 10.1101/2025.07.03.25330855. PMID 40630565
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Elyanow R, Snyder TM, Dalai SC, Gittelman RM, Boonyaratanakornkit J, Wald A, Selke S, Wener MH, Morishima C, Greninger AL, Gale M Jr, Hsiang TY, Jing L, Holbrook MR, Kaplan IM, Zahid HJ, May DH, Carlson JM, Baldo L, Manley T, Robins HS, Koelle DM. T cell receptor sequencing identifies prior SARS-CoV-2 infection and correlates with neutralizing antibodies and disease severity. JCI Insight. 2022 May 23;7(10):e150070. doi: 10.1172/jci.insight.150070. PMID 35439166
- [Derived] Senefeld JW, Johnson PW, Kunze KL, Bloch EM, van Helmond N, Golafshar MA, Klassen SA, Klompas AM, Sexton MA, Diaz Soto JC, Grossman BJ, Tobian AAR, Goel R, Wiggins CC, Bruno KA, van Buskirk CM, Stubbs JR, Winters JL, Casadevall A, Paneth NS, Shaz BH, Petersen MM, Sachais BS, Buras MR, Wieczorek MA, Russoniello B, Dumont LJ, Baker SE, Vassallo RR, Shepherd JRA, Young PP, Verdun NC, Marks P, Haley NR, Rea RF, Katz L, Herasevich V, Waxman DA, Whelan ER, Bergman A, Clayburn AJ, Grabowski MK, Larson KF, Ripoll JG, Andersen KJ, Vogt MNP, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, Buchholtz ZA, Pletsch MC, Wright K, Greenshields JT, Joyner MJ, Wright RS, Carter RE, Fairweather D. Access to and safety of COVID-19 convalescent plasma in the United States Expanded Access Program: A national registry study. PLoS Med. 2021 Dec 20;18(12):e1003872. doi: 10.1371/journal.pmed.1003872. eCollection 2021 Dec. PMID 34928960
- [Derived] Kunze KL, Johnson PW, van Helmond N, Senefeld JW, Petersen MM, Klassen SA, Wiggins CC, Klompas AM, Bruno KA, Mills JR, Theel ES, Buras MR, Golafshar MA, Sexton MA, Diaz Soto JC, Baker SE, Shepherd JRA, Verdun NC, Marks P, Paneth NS, Fairweather D, Wright RS, van Buskirk CM, Winters JL, Stubbs JR, Senese KA, Pletsch MC, Buchholtz ZA, Rea RF, Herasevich V, Whelan ER, Clayburn AJ, Larson KF, Ripoll JG, Andersen KJ, Lesser ER, Vogt MNP, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, Casadevall A, Carter RE, Joyner MJ. Mortality in individuals treated with COVID-19 convalescent plasma varies with the geographic provenance of donors. Nat Commun. 2021 Aug 11;12(1):4864. doi: 10.1038/s41467-021-25113-5. PMID 34381030
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Joyner MJ, Carter RE, Senefeld JW, Klassen SA, Mills JR, Johnson PW, Theel ES, Wiggins CC, Bruno KA, Klompas AM, Lesser ER, Kunze KL, Sexton MA, Diaz Soto JC, Baker SE, Shepherd JRA, van Helmond N, Verdun NC, Marks P, van Buskirk CM, Winters JL, Stubbs JR, Rea RF, Hodge DO, Herasevich V, Whelan ER, Clayburn AJ, Larson KF, Ripoll JG, Andersen KJ, Buras MR, Vogt MNP, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, Paneth NS, Fairweather D, Wright RS, Casadevall A. Convalescent Plasma Antibody Levels and the Risk of Death from Covid-19. N Engl J Med. 2021 Mar 18;384(11):1015-1027. doi: 10.1056/NEJMoa2031893. Epub 2021 Jan 13. PMID 33523609
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747
- [Derived] Joyner MJ, Senefeld JW, Klassen SA, Mills JR, Johnson PW, Theel ES, Wiggins CC, Bruno KA, Klompas AM, Lesser ER, Kunze KL, Sexton MA, Diaz Soto JC, Baker SE, Shepherd JRA, van Helmond N, van Buskirk CM, Winters JL, Stubbs JR, Rea RF, Hodge DO, Herasevich V, Whelan ER, Clayburn AJ, Larson KF, Ripoll JG, Andersen KJ, Buras MR, Vogt MNP, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, Paneth NS, Fairweather D, Wright RS, Carter RE, Casadevall A. Effect of Convalescent Plasma on Mortality among Hospitalized Patients with COVID-19: Initial Three-Month Experience. medRxiv [Preprint]. 2020 Aug 12:2020.08.12.20169359. doi: 10.1101/2020.08.12.20169359. PMID 32817978
- [Derived] Piechotta V, Chai KL, Valk SJ, Doree C, Monsef I, Wood EM, Lamikanra A, Kimber C, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Jul 10;7(7):CD013600. doi: 10.1002/14651858.CD013600.pub2. PMID 32648959
- [Derived] Joyner MJ, Wright RS, Fairweather D, Senefeld JW, Bruno KA, Klassen SA, Carter RE, Klompas AM, Wiggins CC, Shepherd JR, Rea RF, Whelan ER, Clayburn AJ, Spiegel MR, Johnson PW, Lesser ER, Baker SE, Larson KF, Ripoll JG, Andersen KJ, Hodge DO, Kunze KL, Buras MR, Vogt MN, Herasevich V, Dennis JJ, Regimbal RJ, Bauer PR, Blair JE, Van Buskirk CM, Winters JL, Stubbs JR, Paneth NS, Verdun NC, Marks P, Casadevall A. Early safety indicators of COVID-19 convalescent plasma in 5000 patients. J Clin Invest. 2020 Sep 1;130(9):4791-4797. doi: 10.1172/JCI140200. PMID 32525844
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: Expanded Access to Convalescent Plasma for the Treatment of Patients With COVID-19 — http://www.USCOVIDplasma.org